CLINICAL TRIAL: NCT00523887
Title: Post-Marketing Surveillance of Durogesic for Treatment Pain Caused by Radiotherapy
Brief Title: Fentanyl for Treatment Pain Caused by Radiotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013990
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Pain
Keywords: Radiation pain; Duragesic; Fentanyl; Pain
MeSH Terms: conditions — Pain

INTERVENTIONS:
Drug: Fentanyl transdermal therapeutic system

SUMMARY:
The purpose of this study is to assess the clinical utility and safety of Fentanyl for pain treatment caused by radiotherapy. Fentanyl is a synthetic pure opioid agonist with a selective activity on µ receptors.

DETAILED DESCRIPTION:
The study is a phase IV, open label, single arm study. The purpose of this study is to assess the clinical utility and safety of fentanyl transdermal therapeutic system (patch) for treatment of pain caused by radiotherapy. The patients increase or even decrease the amount of study medication in order to achieve pain relief, 48 to 72 hours or 3 days are required after the first patch application. The study medication will be used for 4 weeks. VAS (visual analog scale), BPI Q9 (quality of life) and global assessment have been used to assess the effectiveness. VAS will be assessed every week. BPI Q9 will be assessed at week 1 and week 4. Global assessment will be assessed at week 4. The safety of the study drug will be evaluated using adverse event (AE) report.

The investigator will assess the pain intensity of patients and increase or even decrease Fentanyl dosage every week. Fentanyl will be started on 25 or 50 ug per hr depending on investigator's judgement. Fentanyl will be administered for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients have the history of head and neck tumor
* Patients who are proceeding radiotherapy
* Patients who are administered weak opioids and pain score (Visual analog scale) of 4

Exclusion Criteria:

* Patients who have been administered Fentanyl for pain treatment within 2 weeks before the study
* Patients who will have surgery within 1 month
* Known presence of distant metastasis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2005-08; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical utility of Fentanyl transdermal therapeutic system for pain treatment caused by radiotherapy. VAS (at week 1~4), BPI Q9 (week 1 and 4) and global assessment (week 4) have been used to assess the clinical utility.

SECONDARY OUTCOMES:
To evaluate the safety of Fentanyl transdermal therapeutic system for pain treatment caused by radiotherapy using AE (adverse event) report at every visit.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd